CLINICAL TRIAL: NCT07168681
Title: The Effects of Visual Input on Cognitive Function, Physical Performance, and Postural Stability in Adolescent Male Basketball Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HÜ- FTR- BD- 5
Record Dates: First submitted 2025-08-12; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sports Physical Therapy; Stroboscopic Visual Training; Cognitive Function; Physical Performance; Postural Stability
Keywords: physical performance; stroboscopic visual training; cognitive function
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroboscopic visual training group (Experimental): The exercise program to be implemented within the scope of the study is the SHRed (Sports Injury Prevention for the Lower Extremity, focusing on musculoskeletal and head-related injuries) neuromuscular training program. The program will be administered over six weeks, with two sessions per week. In the experimental group, the exercises will be performed using stroboscopic glasses.
  For the experimental group, the exercises with stroboscopic glasses will be administered in intervals of 2.5 minutes of exercise followed by 2.5 minutes of rest.
  Interventions: Other: Control group
- Control group (Active Comparator): The exercise program to be implemented within the scope of the study is the SHRed (Sports Injury Prevention for the Lower Extremity, focusing on musculoskeletal and head-related injuries) neuromuscular training program. The program will be administered over six weeks, with two sessions per week.
  Participants will be randomly assigned into two groups. The experimental group will perform the exercises while wearing stroboscopic glasses, whereas the control group will perform the exercises under normal visual conditions.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Control group — Active Comparator: Control group The exercise program to be implemented within the scope of the study is the SHRed (Sports Injury Prevention for the Lower Extremity, focusing on musculoskeletal and head-related injuries) neuromuscular training program. The program will be administered over six weeks, with two sessions per week.
  The control group will perform the exercises under normal visual conditions. The exercise program to be implemented within the scope of the study is the SHRed (Sports Injury Prevention for the Lower Extremity, focusing on musculoskeletal and head-related injuries) neuromuscular training program. The program will be administered over six weeks, with two sessions per week. Previous research has shown that the SHRed injury prevention neuromuscular training program reduces ankle and knee injuries in youth basketball players by 36% [35]. The program consists of balance, agility, strength, and aerobic exercises.
  Other Names: Exercise training under normal visual conditions

SUMMARY:
The aim of this study is to investigate the effects of exercises performed with stroboscopic glasses-recently gaining popularity in sports-on cognitive function, physical performance, and postural stability, which are among the key skills in athletic performance.

The originality of the study lies in being the first to examine the effects of stroboscopic glasses-based exercises on basketball players.

Hypotheses of the study:

H1: Exercises performed with stroboscopic glasses have an effect on athletes' cognitive functions.

H2: Exercises performed with stroboscopic glasses have an effect on athletes' physical performance.

H3: Exercises performed with stroboscopic glasses have an effect on athletes' static and dynamic postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players aged 14-19 years
* With at least one year of basketball experience
* Minimum training frequency of two days per week.

Exclusion Criteria:

* Not willing to participate in the study
* A history of any upper or lower extremity surgery within the past year
* A history of any musculoskeletal injury in the upper or lower extremities within the past month
* The presence of a neurological disorder
* A history of epilepsy
* A diagnosis of attention deficit hyperactivity disorder (ADHD)

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Day 1, after the 6 weeks and after the 4 weeks
  It is planned to conduct the assessment using the Central Nervous System Vital Signs test battery. The Central Nervous System Vital Signs is a computer-based neurocognitive test battery with established validity and reliability, and is utilized in 66 countries.

SECONDARY OUTCOMES:
Static Postural stability | Day 1, after the 6 weeks and after the 4 weeks
  Postural stability will be assessed statically using the GYKO inertial sensor. The GYKO inertial sensor system (dimensions: 50 × 70 × 20 mm, weight: 35 g; Microgate, Bolzano, Italy) includes a three-dimensional accelerometer, gyroscope, and magnetometer, enabling data acquisition at a sampling frequency of 500 Hz (full-scale range: 8 g).
Dynamic Postural stability | Day 1, after the 6 weeks and after the 4 weeks
  Dynamic postural stability will be assessed using the Lower Extremity Y Balance Test, which is employed to evaluate dynamic balance, mobility, and neuromuscular control.
Change of direction ability | Day 1, after the 6 weeks and after the 4 weeks
  In the assessment of physical performance, change of direction ability, reactive agility, and jumping performance will be evaluated. The change-of-direction (COD) ability will be assessed using the V-Cut Test. The V-Cut Test is a valid and reliable COD assessment for young basketball players (ICC = 0.92) [26].
  In this test, athletes perform a 25-meter sprint incorporating a 45° change of direction every 5 meters. The total completion time of the test is recorded.
Reactive agility | Day 1, after the 6 weeks and after the 4 weeks
  In the assessment of physical performance, change of direction ability, reactive agility, and jumping performance will be evaluated. Reactive agility assess Y shaped test. The Y-Shaped Agility Test will be administered to evaluate reactive agility performance. This test is specifically designed to represent the change-of-direction movements and running patterns frequently encountered in basketball [29]. The protocol consists of a 5-meter straight sprint followed by a 45° change of direction to either the left or right side, followed by another 5-meter sprint. Athletes begin from a stationary position 30 cm behind the starting line, and timing is initiated once the first photocell gate is crossed. After completing the initial 5-meter sprint, the athlete changes direction to the predetermined side (left or right) and sprints an additional 5 meters. The timing is stopped when the athlete passes through the second photocell gate.
Jumping Performance | Day 1, after the 6 weeks and after the 4 weeks
  In the assessment of physical performance, change of direction ability, reactive agility, and jumping performance will be evaluated. Jump performance will be assessed using the My Jump Lab application.
  Athletes will perform one familiarization trial at submaximal effort, followed by a 1-minute rest period, and then complete three vertical jumps.
  The validity and reliability of the My Jump Lab application have been previously demonstrated.

IPD SHARING:
Plan to Share IPD: No